CLINICAL TRIAL: NCT02140957
Title: Office Based Intervention to Reduce Bottle Use in Toddlers: TARGet Kids! Pragmatic Randomized Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Jonathon Maguire, Staff Physician, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1000032247
Record Dates: First submitted 2013-08-19; First posted 2014-05-16 (Estimated); Results first posted 2016-02-05 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2016-01

CONDITIONS: Educational Intervention and Toddler Bottle Use
Keywords: Toddler Bottle Use; Educational Intervention; Pediatrics; Iron Deficiency
MeSH Terms: conditions — Iron Deficiencies | interventions — Early Intervention, Educational

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Educational Intervention (Experimental): Parents in this arm received a 5 minute educational intervention on bottle cessation plus standard nutritional counseling.
  Interventions: Behavioral: Educational Intervention
- Control (Placebo Comparator): Parents in this arm received a placebo which consisted of standard nutritional counseling alone.
  Interventions: Behavioral: Educational Intervention

INTERVENTIONS:
Behavioral: Educational Intervention — Parents of children in both intervention and control groups received standardized counseling on healthy nutrition based on Canadian Paediatric Society guidelines. In addition, during the same 9-month doctors visit, parents of infants allocated to the intervention group were given a sip cup (Avent Magic CupTM) and shown how to use it. A trained research assistant told intervention group parents the risks of continued bottle use. They were also instructed to limit daily milk consumption to 16 ounces. Parents were also counseled to discontinue bottle use in the next 1 week using a step-wise protocol described on a handout to be placed on their refrigerator. Parents of infants allocated to the control group did not receive this information.

SUMMARY:
Observational studies support an association between bottle feeding beyond 15 to 18 months of age and lower socioeconomic status, excessive milk intake, dental caries, iron deficiency, behavioral issues and obesity. Yet many parents, particularly those from low socioeconomic households, choose to feed their children by bottle much beyond this age. Recognizing the need for further educational interventions for bottle feeding, the TARGet Kids! Research Collaboration recently developed a 5-minute bottle weaning educational intervention for the 9 month well-child visit. We undertook a pragmatic randomized controlled trial to evaluate its effectiveness involving 251 children recruited through TARGet Kids! (PMID: 20624802) The goal was to determine whether an office-based, educational intervention for parents of 9-month-old children could reduce bottle use and iron depletion at 2 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Children and their families who participated in The Applied Research Group for Kids (TARGet Kids!) pragmatic RCT

Exclusion Criteria:

* N/A

Ages: 6 Months to 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 251 (Actual)
Dates: Start 2007-01; Primary Completion 2009-09 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathon Maguire, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Educational Intervention | Control
Started | 129 | 122
Completed | 102 | 99
Not Completed | 27 | 23

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Educational Intervention | Control | Total
Number analyzed (Participants) | 129 | 122 | 251
Age, Continuous [Mean (Standard Deviation); unit: months] | 9.25 (0.38) | 9.24 (0.41) | 9.25 (0.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 53 | 119
  Male | 63 | 69 | 132

OUTCOME MEASURES:

1. Primary Outcome: Change in Iron Depletion
Description: Iron depletion (serum ferritin < 10 μg/L).
Time Frame: Baseline, 2 years
Measure: Number; unit: percentage of participants
Arm/Group | Educational Intervention | Control
Number analyzed (Participants) | 102 | 99
percentage of participants
  Iron depletion - No | 88 | 83
  Iron depletion - Yes | 12 | 17

2. Secondary Outcome: Current Bottle Use
Description: Current daytime bottle use.
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Educational Intervention | Control
Number analyzed (Participants) | 102 | 99
participants | 15 | 40

3. Secondary Outcome: Current Nighttime Bottle Use
Description: Current nighttime bottle use.
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Educational Intervention | Control
Number analyzed (Participants) | 102 | 99
participants | 3 | 10

ADVERSE EVENTS:
Arm/Group | Educational Intervention | Control
Serious Adverse Events (participants affected / at risk) | 0/129 | 0/122
Other Adverse Events (participants affected / at risk) | 0/129 | 0/122

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes